CLINICAL TRIAL: NCT05074472
Title: A Phase 1/2, First-in-Human, Open Label, Dose Escalation Study Of A Cancer-Specific Plectin (CSP)-Targeting Functional Antibody in Solid Tumors That Are Likely to Express CSP
Brief Title: A Phase 1/2, First-in-Human, Open Label, Dose Escalation Study Of A CSP Targeting Functional Antibody in Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ZielBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZIEL-ZB131-101
Record Dates: First submitted 2021-09-23; First posted 2021-10-12 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult; Pancreatic Ductal; Adenocarcinoma; Ovarian Serous Adenocarcinoma; Biliary Cancer Metastatic; Ovarian Serous Cystadenocarcinoma
Keywords: Advanced or Metastatic Ovarian Cancer (ovarian serous adenocarcinoma; ovarian serous cystadenocarcinoma); Advanced or Metastatic Biliary Cancer (intrahepatic, extrahepatic, gallbladder); Advanced or Metastatic Pancreatic Cancer (pancreatic ductal; adenocarcinoma)
MeSH Terms: conditions — Adenocarcinoma; Ovarian Neoplasms; Biliary Tract Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Treatment: ZB131 (Experimental): During the Dose Escalation Stage, patients will be treated with ZB131 at increasing dose levels, beginning with a starting dose level (DL0) of 3 mg/kg once weekly, up to a maximum dose level (DL3) of 15 mg/kg once weekly.
  Interventions: Drug: ZB131

INTERVENTIONS:
Drug: ZB131 — ZB131 will be administered once weekly by intravenous infusion with the weight at baseline used for mg/kg dose calculations.

SUMMARY:
This study is a first-in-human, Phase 1, open label, multicenter, dose escalation study with expansion at the RP2D, to evaluate the safety, tolerability, and preliminary efficacy of ZB131 in patients with solid tumors where prevalence of CSP expression is high. Approximately 12 to 24 patients will be enrolled in the Dose Escalation Stage; the total number of patients will depend on the dose level at which the RP2D is defined. Patients who meet the eligibility criteria during Screening will enter the treatment period. ZB131 will be given via IV every week. Patients will be treated until disease progression or unacceptable toxicities occur.

DETAILED DESCRIPTION:
This study is a first-in-human, Phase 1, open label, multicenter, dose escalation study with expansion at the RP2D, to evaluate the safety, tolerability, and preliminary efficacy of ZB131 in patients with solid tumors where prevalence of CSP expression is high. Approximately 12 to 24 patients will be enrolled in the Dose Escalation Stage; the total number of patients will depend on the dose level at which the RP2D is defined. Patients who meet the eligibility criteria during Screening will enter the treatment period. ZB131 will be given via IV every week. Patients will be treated until disease progression or unacceptable toxicities occur.

Once the RP2D has been established, the Dose Expansion stage will begin to enroll subjects by cohort. For each expansion cohort, subjects will be enrolled in two stages. The first stage includes an evaluation of 12 patients. If 1 or more of 12 patients have a CR or PR, then accrual will continue until a total of 37 patients with measurable disease have been enrolled. Additional patients may be added to ensure 37 subjects with measurable disease are available for evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of signing informed consent.
2. Diagnosis of histologically or cytologically confirmed advanced solid tumors

   1. Dose Escalation Stage: patients with solid tumors (excluding melanoma and hepatocellular CR) who have failed all available therapies or are not eligible for standard of care (SOC).
   2. Dose Expansion Stage:

   i. Cohort A: Advanced or Metastatic Pancreatic Cancer (pancreatic ductal; adenocarcinoma) who have failed or are not eligible for SOC; ii. Cohort B: Advanced or Metastatic Ovarian Cancer of the serous type (ovarian serous adenocarcinoma; ovarian serous cystadenocarcinoma) who have failed or are not eligible for SOC; iii. Cohort C: Advanced or Metastatic Biliary Cancer (intrahepatic, extrahepatic, gallbladder) who have failed or are not eligible for SOC.
3. Eastern Cooperative Oncology Group (ECOG) status of 0-1.
4. Measurable disease per RECIST as assessed by local site investigator/radiologists; lesions situated in previous irradiated areas are considered measurable if progression has been demonstrated in such lesions.
5. Patients must have a tumor lesion that can be safely biopsied and agree to provide a fresh or archival tissue sample prior to treatment initiation and agree to an on-treatment biopsy. The on-treatment biopsy may be waived for patients in the Dose Escalation Stage if a biopsy sample is not possible. An archival sample must be ≤6 months old.
6. Locally advanced, recurrent, or metastatic neoplastic disease that has failed to respond to standard therapy, is not curable by currently available local therapies, or for whom no appropriate therapies are available (based on the judgement of the Investigator.
7. Life expectancy of ≥3 months in the judgement of the Investigator
8. Adequate hematologic function based on the following:

   a. Absolute neutrophil count ≥1.5 x 109/L b. Platelet count ≥100 x 109/L c. Hemoglobin ≥9.0 g/dL
9. Adequate coagulation parameters based on the following:

   a. Prothrombin Time-International Normalized Ratio/partial thromboplastin time (PT-INR/PTT) < ) <1.5 x ULN, unless coumarin derivatives are used; and b. Partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) <1.25 x ULN (therapeutic anticoagulation.

   Note: Anti-coagulation therapy is allowed, if this treatment canpermitted but should be able to be interrupted for a biopsy as judgedif deemed necessary by the Investigator).. The coagulation parameters for patients on anti-coagulation will be interpreted according to expected institutional therapeutic parameters.
10. Adequate hepatic function based on the following:

    a. Total bilirubin <1.5 × upper limit of normal (ULN) (unless elevated due to Gilbert's syndrome [≤3.0 × ULN]) and/or isolated elevations of indirect bilirubin are eligible for study participation; b. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 × ULN for patients with known hepatic metastases).
11. Adequate renal function based on serum creatinine clearance ≥45 mL/min (normal to moderate renal impairment) as determined by Cockcroft-Gault equation may be included in both the Dose Escalation and Dose Expansion stages.
12. Female patients of childbearing potential must have a negative pregnancy test. For women of childbearing potential (WCBP), defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 12 consecutive months for women >55 years of age, a negative serum or urine pregnancy test must be obtained within 72 hours before first treatment. WCBP should be placed on effective birth control directly after testing negative for pregnancy; if not, then WCBP should have a pregnancy test on Day 1 of every dosing cycle, prior to drug administration. Any positive or indeterminant urine pregnancy test (UPT) result must be confirmed by serum pregnancy test.
13. Female patients of childbearing potential must use a highly effective mode of contraception or abstain from heterosexual activity for the duration of the trial and for 120 days following the last dose of study medication. Highly effective contraception includes oral hormonal contraceptives, hormonal contraceptive implant, injection or patch, intrauterine device, or complete abstinence from sexual intercourse.
14. Male patients must agree to use highly effective contraception. Sexually active males who have not had a vasectomy, and whose partner is reproductively capable, must agree to abstain from sexual intercourse or use barrier contraception from Screening through 120 days after their last dose of study treatment.
15. Ability to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Major surgery within 4 weeks prior to Screening. Major surgery is any invasive operative procedure in which a more extensive resection is performed, e.g. a body cavity is entered, organs are removed, or normal anatomy is altered. In general, if a mesenchymal barrier is opened (pleural cavity, peritoneum, meninges), the surgery is considered major. Minimally invasive (laparoscopic) procedures are not considered major surgery, unless considered high risk and requiring extended (greater than over- night observation).
2. Prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids for their radiation therapy, and no history of radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease.
3. Anti-cancer therapy, such as chemotherapy, immunotherapy, hormonal therapy, targeted therapy, or investigational agents within five half-lives or four weeks, whichever is shorter, prior to administration of the first dose of study treatment. Hormonal therapy as maintenance when there is no evaluable cancer is allowed.
4. Active CNS metastases; however, patients who have undergone radiation and/or surgery for the treatment of CNS metastases, who are neurologically stable, and who are no longer taking pharmacologic doses of corticosteroids are eligible; patients with leptomeningeal metastases are not eligible.
5. Primary CNS malignancy.
6. Evidence of metastatic ileus on CT.
7. Severe gastrointestinal conditions such as clinical or radiological evidence of bowel obstruction within 4 weeks prior to study entry;
8. Known active Infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C virus (HCV):

   a. Patients with HIV are excluded.

   a.b. Patients who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment.

   i. Note: Patients should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.

   ii. Hepatitis B screening tests are not required unless:

1. Known history of HBV infection, 2. Mandated by local health authority. b.c. Patients with a history of hepatitis C virus infection are eligible if HCV viral load is undetectable at Screening.

i. Note: Patients must have completed curative antiviral therapy at least 4 weeks prior to enrollment.

ii. Hepatitis C screening tests are not required unless: 1. Known history of HCV infection, 2. Mandated by local health authority. 9. Requiring immunosuppressive therapy. 10. Ongoing systemic bacterial, fungal, or viral infections at Screening;

a. Note: Patients on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met.

11. Received a live vaccine within 6 weeks of first dose of study drug. 12. Received a COVID-19 vaccine less than 1 week prior to dosing (Cycle 1 / Day 1) and/or during the study received a COVID-19 vaccine or booster less than 3 weeks ahead of a tumor assessment.

13. Baseline QT interval corrected with Fridericia's method (QTcF) >480 ms.

a. Note: Criterion does not apply to patients with a right or left bundle branch block.

14. Female patients who are pregnant or breastfeeding. 15. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or prostate intraepithelial neoplasia.

16. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.

17. History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening.

a. Note: Current atrial fibrillation that is on treatment and under control is permitted.

18. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 1 month
  Determine maximum plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, MD, Study Director — ZielBio, Inc.
Locations (9):
- United States (9):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - NEXT Onoology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No